CLINICAL TRIAL: NCT05373758
Title: A Randomized Clinical Trial to Evaluate Solutions for the Management of Virologic Failure for Individuals on Tenofovir, Lamivudine, and Dolutegravir (TLD) in Sub-Saharan Africa
Brief Title: A Randomized Clinical Trial to Evaluate Solutions for the Management of Virologic Failure on TLD in Sub-Saharan Africa
Acronym: RESOLVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mbarara University of Science and Technology (Other); University of KwaZulu (Other); University of California, San Francisco (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Suzanne McCluskey, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022P001193; R01AI167699 (NIH)
Record Dates: First submitted 2022-05-06; First posted 2022-05-13 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: HIV Infections; AIDS; Virologic Failure
Keywords: ART; Medication Adherence; Drug resistance; Dolutegravir
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Standard of Care (Experimental): In Uganda, participants will be managed per Ministry of Health (MOH) guidelines. GRT is performed by MOH for individuals with virologic failure on TLD. Participants will continue enhanced adherence counseling (EAC) and TLD while awaiting the GRT result. Treatment decision will be made by the regional switch committee when GRT results return. There will be a Week 24 visit for specimen collection.
  In South Africa, participants will be managed per Department of Health (DOH) guidelines. Some individuals will be eligible for GRT (performed by DOH) based on ART duration and adherence per DOH guidelines. Treatment decision will be made by the clinic when GRT results return. Individuals who are ineligible for GRT will undergo EAC and continue on TLD. At Weeks 24, participants will undergo plasma HIV-1 RNA viral load testing. Results will be returned to the clinic team for patient management per DOH guidelines.
  All participants undergo viral load testing at Week 48.
  Interventions: Other: Standard of Care treatment strategy
- Individualized Care (Experimental): Participants will undergo routine EAC, point-of-care urine tenofovir (TFV) testing, and genotypic resistance testing (GRT) at enrollment. Participants will return when GRT results are available for a treatment decision. Side effects and tolerance will also be assessed. All information will be used to make an optimal treatment recommendation with participant input. Participants will have an additional study visit at Week 24 and will continue to have routine care visits, adherence counseling by the clinic, and viral load monitoring at intervals determined by the clinic per national guidelines. Participants will undergo plasma HIV-1 RNA viral load testing at Week 48.
  Interventions: Other: Individualized Care treatment strategy
- Immediate Switch (Experimental): Participants will undergo routine EAC and a switch from TLD to PI-based second-line ART at the enrollment visit (Week 0). Participants will have an additional study visit at Week 24. Participants will continue to have routine care visits and viral load monitoring at intervals determined by the clinic per national guidelines. At study completion, participants will undergo plasma HIV-1 RNA viral load testing at Week 48.
  Interventions: Other: Immediate Switch

INTERVENTIONS:
Other: Standard of Care treatment strategy — Management of virologic failure on TLD using the Standard of Care strategy
  Arms: Standard of Care
Other: Individualized Care treatment strategy — Management of virologic failure on TLD using the Individualized Care strategy
  Arms: Individualized Care
Other: Immediate Switch — Management of virologic failure on TLD using the Immediate Switch strategy
  Arms: Immediate Switch

SUMMARY:
The RESOLVE trial is an open, parallel arm, randomized clinical trial which aims to determine the optimal strategy for management of virologic failure on antiretroviral therapy (ART) with tenofovir, lamivudine, and dolutegravir (TLD) in sub-Saharan Africa. The primary outcome of interest will be viral suppression to <50 copies/mL at 48 weeks using the FDA snapshot definition. The study will be conducted in Uganda and South Africa.

DETAILED DESCRIPTION:
The RESOLVE trial is an open, parallel arm, randomized clinical trial which will be conducted at public-sector HIV clinics in Uganda and South Africa. We will enroll individuals with HIV age 15 and above who have had two HIV-1 RNA viral load results >1,000 copies/mL while on TLD and who have been on TLD for at least 12 months. Participants will be randomized using an equal allocation ratio of 1:1:1 across three study arms: a) Standard of Care (regimen guided by genotypic resistance tests and care as per guidelines in Uganda; and with regimen selection and possible genotypic resistance testing (GRT) and care as per guidelines in South Africa), 2) Individualized Care with regimen choice based on results of genotypic resistance tests and urine tenofovir adherence assays, or 3) Immediate Switch to PI-based second-line ART. Randomization will be stratified by clinic, prior exposure to non-nucleoside reverse transcriptase inhibitors, and virologic failure history. We will follow participants for one year with study visits at enrollment, Week 24, and Week 48. The primary outcome of interest will be viral suppression to <50 copies/mL at 48 weeks using the FDA snapshot definition.

ELIGIBILITY:
Inclusion Criteria:

* Age 15 years and above
* Enrolled in HIV care at one of the study clinics
* History of two HIV-1 RNA viral load measurements >1,000 copies/mL while on TLD
* On TLD for at least 12 months
* Lives within 100 kilometers of study clinic

  * Pregnant women are eligible for enrollment.

Exclusion Criteria:

* Plans to transfer out of the clinic within the next 48 weeks
* Plans to move out of the study catchment area within the next 48 weeks
* As determined by chart review, we will exclude those with known virologic failure on protease inhibitors or exposure to integrase strand transfer inhibitors other than dolutegravir.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 648 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Viral suppression at 48 weeks | 48 weeks post-enrollment (visit window spanning 42 to 54 weeks post-enrollment)
  A plasma HIV-1 RNA viral load <50 copies/mL (FDA-snapshot definition)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne McCluskey, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- RK Khan Hospital Clinic, Durban, South Africa
- Uganda (2):
  - Mbarara City Clinic, Mbarara
  - Mbarara Regional Referral Hospital Immune Suppression Syndrome Clinic, Mbarara